CLINICAL TRIAL: NCT00680628
Title: Randomized Trial of Tenecteplase to Treat Severe Submassive Pulmonary Embolism
Brief Title: Clot Dissolving Treatment for Blood Clots in the Lungs
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI changed institution and impossible to solve problem with contract's sites
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-08-01A
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Tenecteplase; Enoxaparin; Thrombosis; Fibrinolytics
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis | interventions — Tenecteplase; Enoxaparin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Saline + Enoxaparin
  Interventions: Drug: 0.9% Saline + Enoxaparin
- 1 (Experimental): Tenecteplase + Enoxaparin
  Interventions: Drug: Tenecteplase + Enoxaparin

INTERVENTIONS:
Drug: Tenecteplase + Enoxaparin — Enoxaparin: 1 mg/kg within 12 hours before receiving tenecteplase.Subsequently, patients will receive 1 mg/kg enoxaparin SQ Q12 hours until discontinuation is clinically indicated.
  Tenecteplase:will be administered using a tiered-dosing schedule according to patient weight: <60Kg=30mg; ≥60Kg to <70Kg=35mg; ≥70Kg to <80Kg=40mg; ≥80Kg to <90Kg=45mg; ≥90Kg=50mg
  Arms: 1
Drug: 0.9% Saline + Enoxaparin — Enoxaparin: 1 mg/kg within 12 hours before receiving saline.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if tenecteplase plus enoxaparin is safe and effective in the treatment of patients with severe submassive pulmonary embolism.

DETAILED DESCRIPTION:
This project is a phase III, six-center, randomized trial of tenecteplase to treat severe submassive (systolic blood pressure >90 mm Hg) pulmonary embolism (PE). "Severe" requires one of the following predictors of a adverse outcome: right ventricular (RV) hypokinesis on echocardiography, hypoxemia (pulse oximetry reading <95%, <1000 feet above sea level), serum troponin I (abnormal at local threshold) or brain natriuretic peptide concentration >90 pg/mL (or NT proBNP >900 pg/mL). Patients from the emergency department or inpatients can be enrolled within 24 hours of a diagnostic positive CT angiography. After informed consent, eligible patients will be randomized to the study or placebo arm. All patients will a receive a 1mg/kg enoxaparin, SQ followed by a syringe prepared in pharmacy containing either a body weight-adjusted dose of tenecteplase or a 0.9% saline placebo, given IV push. Patients will be followed for five days post-treatment for composite acute adverse outcomes: PE-related (death, any ACLS intervention, circulatory shock, respiratory failure, need for vasopressors with organ dysfunction) and hemorrhage-related (intracranial or intraspinal hemorrhage and any other hemorrhage requiring transfusion, surgical or endoscopic intervention or a hemostatic drug). Survivors will return at three months for assessment of a delayed adverse outcomes of death or cardiopulmonary functional limitation (CFL): interval medical care for dyspnea + RV dysfunction or pulmonary hypertension on echo + either a NYHA score ≥3 or a 6 minute walk distance <330 m. Together, the acute and delayed outcomes represent composite serious adverse outcomes (SAOs). We hypothesize an absolute 20% reduction in composite serious adverse outcomes in the study arm compared with the placebo arm. The six hospitals represent geographic diversity: Boston, Charlotte, Chicago, Denver, New Haven, and Springfield, MA. To help maintain balance between sites, the six sites will each enroll a maximum of 40 patients until the sample size of N=200 is reached, which allows the 20% effect size to be tested at α =0.05 and β=0.20 with 15% loss to follow-up. The study will employ an intent-to treat analysis. Secondary endpoints include recurrent venous thromboembolism within three months, scores from two validated quality of life questionnaire (VEINES-QOL and SF-36TM) at three months. Human subject safety include requirement that a study MD verify the presence of all inclusion and absence of exclusions in real-time, a method to allow unblinding to the clinical care team, an independent DSMB that will perform 6 interim analyses and will enforce predefined stopping criteria for either safety or efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary vascular imaging positive for PE within the previous 24 hours
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age >17 years
* Evidence of severe PE: RV hypokinesis on echocardiography, abnormal troponin I or T (any non-normal including indeterminate values, using local reference thresholds) or BNP measurement >90 pg/mL or NT proBNP >900 pg/ml (not more than 6 hours prior to CT angiography and not more than 30 hours before enrollment) or a pulse oximetry reading <95% within previous two hours (<93% in Denver).

Exclusion Criteria:

* Systolic blood pressure < 90 mm Hg at time of informed consent
* Do not resuscitate or do not intubate order
* Systemic fibrinolytic treatment within previous 7 days
* Inability to follow-up at 3 months
* Documented gastrointestinal bleeding within previous 30 days
* Active hemorrhage in any of the following sites at the time of enrollment: intraperitoneal, retroperitoneal, pulmonary, uterine, bladder, or nose.
* Head trauma causing loss of consciousness within previous 7 days
* Any history of hemorrhagic stroke
* Ischemic stroke within the past year
* Prior history of heparin-induced thrombocytopenia
* History of intraocular hemorrhage
* Intracranial metastasis
* Known inherited bleeding disorder, e.g., hemophilia
* Platelet count < 50,000/uL
* Prothrombin time with an INR >1.7
* Chest, abdominal, intracranial or spinal surgery within the previous 14 days
* Subacute bacterial endocarditis
* Pregnancy (positive pregnancy test)
* Prior enrollment in the study
* Current treatment with fondiparinux, dalteparin, a direct thrombin inhibitor or administration of a glycoprotein inhibitor within the previous 48 hours.
* Known pericarditis
* Allergy to heparins,or tenecteplase
* Elapsed time that would preclude drug or placebo administration within 24 hours after diagnosis
* Evidence of non-end stage kidney injury (creatinine clearance < 30 ml/min without chronic hemodialysis treatment; chronic hemodialysis-treated patients are eligible)
* Preexisting end-stage cardiopulmonary disease (heart failure with left ventricular ejection fraction <20%, known severe pulmonary hypertension or other lung disease causing permanent dependence upon oxygen)
* Any other condition that the investigator believes would pose a significant hazard to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Kline, MD, Principal Investigator — Carolinas Medical Center
Locations (7):
- United States (7):
  - University of California, Davis Medical Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Carolinas Medical Center, Charlotte, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Utah Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Zuo Z, Yue J, Dong BR, Wu T, Liu GJ, Hao Q. Thrombolytic therapy for pulmonary embolism. Cochrane Database Syst Rev. 2021 Apr 15;4(4):CD004437. doi: 10.1002/14651858.CD004437.pub6. PMID 33857326
- [Derived] Stewart LK, Peitz GW, Nordenholz KE, Courtney DM, Kabrhel C, Jones AE, Rondina MT, Diercks DB, Klinger JR, Kline JA. Contribution of fibrinolysis to the physical component summary of the SF-36 after acute submassive pulmonary embolism. J Thromb Thrombolysis. 2015 Aug;40(2):161-6. doi: 10.1007/s11239-014-1155-5. PMID 25433511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from 8 hospitals from August 2008 until October, 2012. Genentech funded the study. Carolinas Medical Center was the prime contractor site and subcontracted 7 other hospitals.
Pre-assignment Details: The investigator relocated to a new institution in July 2012, which led to insoluble problems with the subcontracts that forced early study closure.
Groups:
- Placebo: Tenecteplase + Enoxaparin
  Tenecteplase + Enoxaparin : Enoxaparin: 1 mg/kg within 12 hours before receiving tenecteplase.Subsequently, patients will receive 1 mg/kg enoxaparin SQ Q12 hours until discontinuation is clinically indicated.
  Tenecteplase:will be administered using a tiered-dosing schedule according to patient weight: <60Kg=30mg; ≥60Kg to <70Kg=35mg; ≥70Kg to <80Kg=40mg; ≥80Kg to <90Kg=45mg; ≥90Kg=50mg
- Tenecteplase: Saline + Enoxaparin
  0.9% Saline + Enoxaparin : Enoxaparin: 1 mg/kg within 12 hours before receiving saline.
Period: Overall Study
Arm/Group | Placebo | Tenecteplase
Started | 43 | 40
Completed | 43 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: see manuscript
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tenecteplase | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 34 | 71
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (14) | 57 (14) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 24 | 20 | 44
Region of Enrollment [Number; unit: participants]
  United States | 43 | 40 | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Cardiogenic Shock or Respiratory Failure From Pulmonary Embolism and Number of Patietnts With Major Hemorrhage
Time Frame: 1,2,3,4, and 5 days
Measure: Number; unit: participants
Arm/Group | Placebo | Tenecteplase
Number analyzed (Participants) | 43 | 40
participants | 1 | 1

2. Primary Outcome: Number With Functional Cardiopulmonary Limitations Assessed With a Composite Measurement (Six Minute Walk Distance, Right Ventricular Function and Quality of Life Score on the SF-36)
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Placebo | Tenecteplase
Number analyzed (Participants) | 43 | 40
participants | 8 | 4

3. Primary Outcome: Number With Recurrent Venous Thromboembolism and/or Severe Post-phlebitic Syndrome
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Placebo | Tenecteplase
Number analyzed (Participants) | 43 | 40
participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Tenecteplase
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/40
Other Adverse Events (participants affected / at risk) | 0/43 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Tenecteplase (N=40)
intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) — led to death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days